CLINICAL TRIAL: NCT05391958
Title: Pharmacodynamics of Injection of Cisatracurium Base on Lean Body Mass Pattern to Maintain Deep Neuromuscular Blockade in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 070733
Record Dates: First submitted 2022-05-07; First posted 2022-05-26 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obese Patients; Laparoscopic Colorectal Surgery
Keywords: Laparoscopy; Cisatracurium; Obesity; Neuromuscular Blockade; Pneumoperitoneum; Pharmacology
MeSH Terms: conditions — Obesity; Pneumoperitoneum | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal Real group (Sham Comparator): the medication group was given according to the actual weight of normal weight patients
  Interventions: Behavioral: base on Actual Body Weight; Genetic: normal patients
- Normal Lean group (Active Comparator): For normal weight patients, the medication group was given according to the lean body mass
  Interventions: Behavioral: base on Lean Body Mass Pattern; Genetic: normal patients
- Obese Real group (Sham Comparator): the medication group was given according to the actual weight of obese weight patients
  Interventions: Behavioral: base on Actual Body Weight; Genetic: obese patients
- Obese Lean group (Experimental): the medication group was given according to the lean body mass of obese weight patients
  Interventions: Behavioral: base on Lean Body Mass Pattern; Genetic: obese patients

INTERVENTIONS:
Behavioral: base on Lean Body Mass Pattern — PTC(post-tetanic count) was measured every 6min during the operation, and single injection of 0.05 (1ED95) mg/kg cisatracurium that was calculated based on lean body weight mass pattern once when PTC > 2.
  Other Names: general anesthesia
  Arms: Normal Lean group; Obese Lean group
Behavioral: base on Actual Body Weight — PTC was measured every 6min during the operation, and single injection of 0.05 (1ED95) mg/kg cisatracurium that was calculated based on actual body weight once when PTC > 2.
  Other Names: base on Actual Body Mass Pattern
  Arms: Normal Real group; Obese Real group
Genetic: obese patients — obese patients with elective laparoscopic colorectal surgery were selected，and the inclusion criteria were as follows: age 18-65, body mass index (BMI) 30-35, waist circumference (WC) : female ≥80cm, male ≥90cm, and American Society of Anesthesiologists (ASA) grade Ⅰ ~ Ⅲ.
  Other Names: laparoscopic colorectal surgery
  Arms: Obese Lean group; Obese Real group
Genetic: normal patients — normal patients with elective laparoscopic colorectal surgery whose body mass index (BMI) 18-24 were selected,and American Society of Anesthesiologists (ASA) grade Ⅰ ~ Ⅲ.
  Other Names: laparoscopic colorectal surgery
  Arms: Normal Lean group; Normal Real group

SUMMARY:
To observe the pharmacodynamics of intravenous injection of cisatracurium to maintain deep neuromuscular blockade in obese patients with lean body mass in laparoscopic colorectal surgery

DETAILED DESCRIPTION:
According to the random number table method, one hundred and twenty patients who underwent elective laparoscopic colorectal surgery were divided into four groups (n=30): Normal weight patients according to lean body weight group(NL group), normal weight patients according to real weight group (NR group), obese patients according to lean body weight group(OL group), and obese patients according to real weight group(OR group).Intraoperative deep neuromuscular blockade (PTC≤2)was maintained in all four groups.The dosage of cisatracurium, the number of injections,time to effect,time to recovery from TOFr,time to recover TOFr（train-of-four rate） to 0.7 and 0.9,and time to stay in PCAU were recorded.The surgeon's satisfaction with the operative field and the average intraoperative pneumoperitoneum pressure were recorded at the time of pneumoperitoneum establishment,1 hour and 2 hours after pneumoperitoneum establishment.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Colorectal Surgery
* American Society of Anesthesiologists (ASA) grades I-III

Exclusion Criteria:

* Patients with heart, lung and other vital organ disorders
* Preoperative fluid and electrolyte disturbance
* Preoperative water and electrolyte disorders have a history of neuromuscular disease or take medications that have an impact on neuromuscular function
* There is a significant airway difficulty
* Refuse to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Change in average dosing interval time | during the surgery
  PTC(post-tetanic count)was measured every 6min during the operation, and cisatracurium was injected once when PTC > 2,average dosing interval time was recorded
Change in Times of adding cisatracurium | during the surgery
  PTC was measured every 6min during the operation, and cisatracurium was injected once when PTC > 2,and recording the total times of injection.
Change in total dosage of cisatracurium | during the surgery
  PTC(post-tetanic count) was measured every 6min during the operation, and cisatracurium was injected once when PTC > 2,and recording the total dosage of total dosage of cisatracurium
Change in time of onset | through study completion, an average of 3 minute after induction
  0.15mg/kg (3ED95) cisatracurium was given to all groups according to actual body weight as induction dose. Tracheal intubation was performed in all groups when TOFr(train of four ratio)=0.recording the time during this process.
Change in TOF(train of four) recovered to 0.7 and 0.9 from the last injection | up to 1 hour after the surgery
  The recovery of TOF(train of four) was continue observed after surgery.Recording the time both when TOF(train of four) recovered to 0.7 and 0.9
Change in time during PACU(postanesthesia care unit) | up to 2 hour after the surgery
  recoding the duration of stay in PACU(postanesthesia care unit)
surgical rating scale(SRS) | during the surgery
  Surgical rating Scale (SRS) was evaluated by surgical surgeons at the beginning, 1h and 2h of surgery, with a range of 1 to 5, corresponding to "extremely poor", "poor", "adequate", "good" and "best".

SECONDARY OUTCOMES:
The change of MAP (mean arterial pressure) | immediately , 10 minutes , 20 minutes , 30 minutes and 40 min later after the first injection
  Mean arterial pressure were recorded immediately , 10 minutes , 20 minutes , 30 minutes , and 40 minutes later after the first injection
The change of HR(heart rate) | immediately , 10 minutes , 20 minutes , 30 minutes and 40 min later after the first injection
  the heart rate were recorded immediately , 10 minutes , 20 minutes , 30 minutes , and 40 minutes later after the first injection
Change in PaCO2 before and after pneumoperitoneum | before and after pneumoperitoneum during the surgery
  arterial blood gas(ABG) was measured before and after pneumoperitoneum.Recording PaCO2 before and after pneumoperitoneum
Incidence of postoperative pain | Immediately after surgery and One day after surgery
  Incidence of postoperative pain (shoulder, lumbar abdomen, arm)
Whether hypoxemia occurs after extubation | within 10 minutes after extubation
  Observe the occurrence of hypoxemia after extubation

CONTACTS AND LOCATIONS:
Overall Officials: PI qinshuang liu, master, Study Director — The First hosptial of Qinhuangdao; yuli guo, master, Study Chair — The First hosptial of Qinhuangdao
Locations (1):
- The First hosptial of Qinhuangdao, Qinhuangdao, China

IPD SHARING:
Plan to Share IPD: No